CLINICAL TRIAL: NCT01720693
Title: A Pilot Study to Examine a Novel Controlled Hypo-Perfusion Technique in Partial Nephrectomy
Brief Title: Novel Controlled Hypo-Perfusion Technique in Partial Nephrectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Hypoperfusion
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Partial Nephrectomy; Renal Cell Carcinoma
Keywords: partial nephrectomy; hypoperfusion; renal function
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hypoperfusion (Experimental): Hypoperfusion of the renal artery
  Interventions: Procedure: Hypoperfusion of renal artery

INTERVENTIONS:
Procedure: Hypoperfusion of renal artery — The renal artery is occluded to 30% of it's baseline, prior to kidney tumour removal

SUMMARY:
Many patients who are candidates for nephron-sparing surgery, partial nephrectomy is now the standard treatment with a surgical, small, clinical T1 tumor (<7 cm). In many recent studies, partial nephrectomy provides equivalent oncologic, and superior functional, outcomes compared with the standard radical nephrectomy over the short and long term (2, 3). Partial nephrectomy techniques, whether open, laparoscopic or robotic, typically involve hilar clamping, which creates the desired bloodless operative field, allowing for more precise tumor excision and renal reconstruction. This hilar clamping eventually may lead to ischemic kidney injury which can compromise the functional outcomes of the remaining kidney.We are working now to develop a novel technique of Hypo-Perfusion by achieving partial renal arterial clamping, with the goal of completely eliminating surgical ischemia to the renal remnant.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years old scheduled for open partial nephrectomy

Exclusion Criteria:

* No prior diagnosis of renal artery disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To perfect the Renal Hypoperfusion during partial nephrectomy is feasible safe and result in better renal function than complete occlusion of renal blood flow | up to 2 weeks prior to surgery and up to 24 hrs post surgery
  renal function will be measured using creatinine, eGFR, 24 hr creat clearance, and NGAL biomarker of acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jewett, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada